CLINICAL TRIAL: NCT06359223
Title: Effect of Coffee Consumption on Postoperative Pain and Intestinal Motility After Caesarean Section: Randomized Controlled Study
Brief Title: Effect of Coffee Consumption on Pain and Intestinal Motility After Caesarean Section:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: KTO Karatay University (Other)
Responsible Party: Principal Investigator, HÜMEYRA YÜKSEL, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2400602
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Operation; Cesarean Section
Keywords: Caesarean Section; Coffee; pain; Motility
MeSH Terms: conditions — Pain | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine group (Experimental): Participants in the intervention group will receive 100 mg caffeine in coffee at 6 and 12 hours after surgery in addition to routine postoperative care. The control group will receive only routine postoperative care. Pain will be assessed using Visual Analog Scale (VAS) and bowel activity will be monitored by time to first defecation, gas passage and bowel sounds.
  Interventions: Dietary Supplement: coffee consumption
- control group (Active Comparator): The control group will receive only routine postoperative care. Pain will be assessed using Visual Analog Scale (VAS) and bowel activity will be monitored by time to first defecation, gas passage and bowel sounds.
  Interventions: Other: control group

INTERVENTIONS:
Dietary Supplement: coffee consumption — After cesarean section, patients will be allowed to drink coffee.
  Arms: caffeine group
Other: control group — Patients will undergo a routine surgical procedure.
  Arms: control group

SUMMARY:
Objective The aim of this study was to investigate whether postoperative coffee intake affects pain levels and bowel motility in women undergoing cesarean delivery.

Design: It will be conducted as a randomized controlled experimental study. Method: It is a randomized controlled experimental study: This randomized controlled clinical trial will be conducted between May and December 2024 in accordance with the Consolidated Standards of Reporting Trials. A total of 60 women will be randomly assigned to the intervention group (n=30) or the control group (n=30). Participants in the intervention group will receive 100 mg caffeine in coffee at 6 and 12 hours after surgery in addition to routine postoperative care. The control group will receive only routine postoperative care. Pain will be assessed using Visual Analog Scale (VAS) and bowel activity will be monitored by time to first defecation, gas passage and bowel sounds.

Keywords: Caesarean section, Coffee, Pain, Motility

ELIGIBILITY:
Inclusion Criteria:

* had a cesarean delivery with spinal anesthesia,
* had a postoperative pain level of 4 or higher,
* could read and write Turkish,
* could communicate effectively with the researchers.

Exclusion Criteria:

* Those who underwent emergency cesarean section,
* Those with pregnancy complications (e.g., preeclampsia, gestational diabetes, placenta previa),
* Those with a history of chronic gastrointestinal disease (e.g., irritable bowel syndrome, Crohn's disease, ulcerative colitis),
* Those with caffeine sensitivity or allergy,
* Those with chronic pain syndrome or analgesic dependence,
* Those who regularly consume coffee (≥2 cups per day),
* Those who experienced intraoperative complications (e.g., bowel or bladder injury),
* Those who could not comply with the study protocol.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 6 hour
  The visual analog scale (VAS ) is a scale with different names at both ends on a 10 cm long vertical or horizon line. In this study, evaluation was made as "0 = no pain" and "10 = the most severe pain".
intestinal motility | 24 hour
  24 hour. The patient's bowel sounds will be listened to during the hours

CONTACTS AND LOCATIONS:
Overall Officials: HÜMEYRA YÜKSEL, Phd, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay Unıversty, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data of the study can be shared by researchers with permission.

REFERENCES:
- [Background] Zamanabadi MN, Alizadeh R, Gholami F, Seyed Mehdi SA, Aryafar M. Effect of caffeine on postoperative bowel movement and defecation after cesarean section. Ann Med Surg (Lond). 2021 Aug 6;68:102674. doi: 10.1016/j.amsu.2021.102674. eCollection 2021 Aug. PMID 34401138
- [Background] Abadi F, Shahabinejad M, Abadi F, Kazemi M. Effect of Acupressure on Symptoms of Postoperative Ileus After Cesarean Section. J Acupunct Meridian Stud. 2017 Apr;10(2):114-119. doi: 10.1016/j.jams.2016.11.008. Epub 2016 Dec 27. PMID 28483182
- [Background] undefined
- [Result] Goymen, A., Simsek, Y., Ozkaplan, S. E., Ozdurak, H. I., Akpak, Y. K., Semiz, A., & Oral, S. (2017). Effect of gum chewing and coffee consumption on intestinal motility in caesarean sections.
- [Result] Tian YT. 2017. China is not"The World's First Cesarean Section Rate".Beijing: Guangming Daily.
- [Result] Curran EA, Khashan AS, Dalman C, Kenny LC, Cryan JF, Dinan TG, Kearney PM. Obstetric mode of delivery and attention-deficit/hyperactivity disorder: a sibling-matched study. Int J Epidemiol. 2016 Apr;45(2):532-42. doi: 10.1093/ije/dyw001. Epub 2016 Apr 10. PMID 27063604
- [Result] Khadem N, Khadivzadeh T. The intelligence quotient of school aged children delivered by cesarean section and vaginal delivery. Iran J Nurs Midwifery Res. 2010 Summer;15(3):135-40. PMID 21589777
- [Result] Souza JP, Betran AP, Dumont A, de Mucio B, Gibbs Pickens CM, Deneux-Tharaux C, Ortiz-Panozo E, Sullivan E, Ota E, Togoobaatar G, Carroli G, Knight H, Zhang J, Cecatti JG, Vogel JP, Jayaratne K, Leal MC, Gissler M, Morisaki N, Lack N, Oladapo OT, Tuncalp O, Lumbiganon P, Mori R, Quintana S, Costa Passos AD, Marcolin AC, Zongo A, Blondel B, Hernandez B, Hogue CJ, Prunet C, Landman C, Ochir C, Cuesta C, Pileggi-Castro C, Walker D, Alves D, Abalos E, Moises E, Vieira EM, Duarte G, Perdona G, Gurol-Urganci I, Takahiko K, Moscovici L, Campodonico L, Oliveira-Ciabati L, Laopaiboon M, Danansuriya M, Nakamura-Pereira M, Costa ML, Torloni MR, Kramer MR, Borges P, Olkhanud PB, Perez-Cuevas R, Agampodi SB, Mittal S, Serruya S, Bataglia V, Li Z, Temmerman M, Gulmezoglu AM. A global reference for caesarean section rates (C-Model): a multicountry cross-sectional study. BJOG. 2016 Feb;123(3):427-36. doi: 10.1111/1471-0528.13509. Epub 2015 Aug 10. PMID 26259689
- [Derived] Tuzmen HD, Yuksel H, Yazar M, Sayar S, Horasanli JE. The effect of coffee consumption on postoperative pain and bowel motility following cesarean section: a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2025 Nov;314:114723. doi: 10.1016/j.ejogrb.2025.114723. Epub 2025 Sep 13. PMID 40967073